CLINICAL TRIAL: NCT04262284
Title: Respreeza® Self-administration and Learning Program (AmAREtTI Study- Auto-Administration de Respreeza® et Programme d'apprenTIssage)
Brief Title: Respreeza® Self-administration and Learning Program (AmAREtTI Study)
Acronym: AmAREtTI
Status: Completed | Type: Observational
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Other Study IDs: AmAREtTI; 2018-A02601-54 (Other: ANSM)
Record Dates: First submitted 2020-02-04; First posted 2020-02-10 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Alpha-1 Antitrypsin Deficiency
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
According to the Respreeza® Summary of Product Characteristics, the initial infusions must be administered under the supervision of a health professional experienced in the treatment of alpha-1 antitrypsin deficiency, although subsequent infusions may be administered at home by the person responsible for care or by the patient.

Clinical data on self-administration of Respreeza® are however limited and the grounds for self-administration are left to the assessment of the attending physician, who needs to ensure that appropriate training is delivered.

In this context, CSL Behring would like to run a clinical study in order to assess the effectiveness of a home self-administration learning program in terms of switching to self-administration, and the long term maintenance of this administration.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥18 years old).
* Patients suffering from AATD treated by Respreeza® through a peripheral vein at home for at least 3 month (consecutives or not). The 3-month period of treatment with Respreeza® does not necessarily correspond to the 3 months prior to inclusion.
* Patient accompanied by a third person at home
* Patients deemed to be suitable by the investigator for self-administration.
* Patients with a life expectancy of over 3 years.
* Patients who have been informed verbally and in writing via the information leaflet and who have signed the informed consent form.

Exclusion Criteria:

- In order to reflect the reality of everyday practice, no non-inclusion criteria are intended except for patient refusal to take part in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from alpha-1 antitrypsin deficiency (AATD) treated by Respreeza®
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2019-10-18 (Actual); Primary Completion 2024-05-06 (Actual); Study Completion 2024-05-06 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who switch to self-administration without the presence of a nurse at the end of the learning program | Up to 8 weeks
  A patient will be permitted to switch to self-administration without the presence of a nurse if the following conditions are met:
  * Three consecutive successful self-administrations by the patient in the presence of the nurse but without assistance during the learning phase.
  * Validation of the learning grid The percentage is based on number of patient switching to self-administration and remains in self-administration 12 months after
Percentage of patients who switch to self-administration without the presence of a nurse | Up to 12 months

SECONDARY OUTCOMES:
Percentage of patients who switch to self-administration without the presence of a nurse | Up to 8 weeks
  A patient will be permitted to switch to self-administration without the presence of a nurse if the following conditions are met:
  * Three consecutive successful self-administrations by the patient in the presence of the nurse but without assistance during the learning phase.
  * Validation of the learning grid The percentage is based on number of patient switching to self-administration
Patient characteristics | At inclusion
  Socio-demographic data, disease history, concomitant treatments, substitution protocol, percentage of theoretical forced expiratory volume at one second (FEV1), diffusing capacity of lung for carbon monoxide (DLCO), distance from home to hospital, type of follow-up (in hospital, in surgery)
Degree of autonomy | At inclusion and 12 months after self-administration
  The change in the degree of autonomy will be defined as the difference between the autonomy assessed at 12 months and inclusion according to an EVA
The time frame for autonomy | Up to 12 months
  The time to achieve autonomy will be defined by the time between the first learning session for self-administration and the first self-administration without nurse.
Evolution of patients Quality of Life with Saint George's Respiratory Questionnaire (SGRQ) | Up to 12 months
Patients satisfaction for treatment administration by a nurse and for self-administration | Up to 12 months
  Satisfaction for treatment administration by a nurse will be assessed at inclusion by visual analog scale (VAS) Satisfaction for self-administration will be assessed after 12 months after the 1st self-administration or in case of study withdrawal by VAS
Satisfaction about learning program | Up to 8 weeks
  Satisfaction about learning program will be assessed at the end of the learning program by VAS
Tolerance and safety | Up to 12 months
  General and local tolerance at the administration site assessed by the nature and number of adverse events (AEs) and immunoglobulin E impaired gas exchange (IGEs).
Compliance/Observance | Up to 8 weeks
  Compliance/observance measured by the number of scheduled and unrealized sessions.
Determining factors for switch to self-administration | Up to 8 weeks
  Determining factors that may be associated with the transition to self-administration (demographics, disease history, concomitant treatments, substitution protocol, FEV1, QoL at inclusion, duration of learning program).

CONTACTS AND LOCATIONS:
Overall Officials: Study Physician, Study Director — CSL Behring SA
Locations (11):
- France (11):
  - CHU Angers, Angers
  - CHU Bordeaux - Hôpital Haut-Lévèque, Bordeaux
  - CHU Grenoble-Alpes, Grenoble
  - CHU Lille, Lille
  - Hospices Civils de Lyon, Lyon
  - Hôpital Saint Joseph, Marseille
  - Hôpital Bichat-Claude-Bernard, Paris
  - CHU Rennes - Hôpital Pontchaillou, Rennes
  - CHU Strasbourg, Strasbourg
  - CHRU Tours, Tours
  - CHU Nancy Brabois, Vandœuvre-lès-Nancy